CLINICAL TRIAL: NCT03246282
Title: A Polychromatic Light Emitting Diode System to Deliver Low Dose Light Directly Into a Peripheral Intravascular Catheter: A Pain Reduction Study
Brief Title: Feasibility of Polychromatic Light Emitting Diode System to Reduce Pain
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: John W. Reeves, MD (Other)
Collaborators: White Clover Research Foundation (Other); White Clover Wellness and Research Center (Unknown)
Responsible Party: Sponsor-Investigator, John W. Reeves, MD, John W. Reeves, MD, White Clover Research Foundation
Organization: White Clover Research Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UVL_P001
Record Dates: First submitted 2017-08-06; First posted 2017-08-11 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution; Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Polychromatic light emitting diode system is a non-significant risk device that administers low-dose light generated by light emitting diode(s). A small adapter attaches directly to a standard 20-guage catheter that threads a small fiber optic through the distal end of the catheter. The optic terminates at the proximal end of the catheter. Polychromatic light is emitted to illuminate the catheter near the site of catheter entrance. Concurrently, normal saline flows through the optic adapter, into and through the 20-gauge catheter.
  Device: UVL1000 Treatment Station Drug: Normal Saline 0.9% Infusion Solution Bag Device: Peripheral Catheterization
  Interventions: Device: UVL1000 Treatment Station; Drug: Normal Saline 0.9% Infusion Solution Bag; Device: Peripheral Catheterization

INTERVENTIONS:
Device: UVL1000 Treatment Station — Non-coherent light source administered 365 nm, 630 nm, and 530 nm at an output intensity of 0.1 mW directly into an existing intravascular 20 gauge 1.0" catheter
Drug: Normal Saline 0.9% Infusion Solution Bag — 250 ml of 0.9% Sodium Chloride Solution
  Other Names: Normal Saline
Device: Peripheral Catheterization — 20-gauge 1.0" catheter

SUMMARY:
This study uses a prospective non-randomized, non-controlled design. One Hundred Fifty (150) subjects presenting with pain will be enrolled into a single treatment group The purpose of the study is to evaluate the feasibility of PLEDS for PIV catheter light delivery for pain reduction, through change between baseline average pain and final average VAS score. The absence of a control group is based on the following reason: The purpose of this investigation is to further the understanding of the feasibility of PLEDS for PIV catheter light delivery for pain management. Further, the results of this investigation will be used (internally only) to determine if subject-perceived reductions in pain warrant proceeding with more controlled, targeted and possibly randomized studies.

DETAILED DESCRIPTION:
This study uses a prospective non-randomized, non-controlled design. One Hundred Fifty (150) subjects presenting with pain will be enrolled into a single treatment group The purpose of the study is to evaluate the feasibility of Polychromatic Light Emitting Diode System (PLEDS) for Peripheral Intravenous (PIV) catheter light delivery for pain reduction, through change between baseline average pain and final average VAS score. The absence of a control group is based on the following reason: The purpose of this investigation is to further the understanding of the feasibility of PLEDS for PIV catheter light delivery for pain management. Further, the results of this investigation will be used (internally only) to determine if subject-perceived reductions in pain warrant proceeding with more controlled, targeted and possibly randomized studies.

PIV therapy has been used for decades as an effective therapy to maintain proper hydration and electrolyte levels. Additionally, PIV therapy can be infused with various agents, including supplements and pharmacological agents. Low-energy light therapy has been established as an alternative treatment for a myriad of medical conditions including reduction of pain. The concurrent administration of low-light therapy and PIV therapy may serve as a viable therapy for the treatment of pain associated with various medical conditions. Accordingly, this study is designed to assess the feasibility of low light therapy via PLEDS integrated into a standard PIV catheter for the purposes of reduction of pain.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form (see Informed Consent Forms)
* Ages 18-70
* Non-Pregnant Female Participants
* Self-reported perceived pain score via "Brief Pain Inventory - Short Form" score of 2 or more.
* No breastfeeding for 1 week prior to enrollment
* Birth control measures to be used throughout the duration of the study for women of child bearing potential
* Powerful antioxidants (e.g. oral antioxidants, Vitamin C and E, glutathione or Myer's cocktail IV infusion therapy) will not be used on treatment days

Exclusion Criteria:

* Active infection along potential intravenous catheter sites
* Use of anti-inflammatory medications on day of treatment and no more than 400mg per day for over 30 days
* Suffering from blood clotting disorders (hypercoagulable condition, thrombocytosis, etc.)
* Participated in a clinical study in the last 14 days
* Breastfeeding
* Currently taking photosensitizing agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The use of polychromatic light therapy delivered through an intravascular catheter to assess the change in self-reported VAS pain score. | 2 weeks
  To evaluate the feasibility of PLEDS for PIV catheter light delivery for the purposes of pain reduction, through assessing the change between baseline average pain (via "Brief Pain Inventory - Short Form") and final average VAS score (via the "Per Treatment VAS Score Form") following treatment administration.

OTHER OUTCOMES:
Subject Satisfaction | 2 weeks
  Self-reported overall treatment satisfaction based on perceived response from treatment

CONTACTS AND LOCATIONS:
Overall Officials: John W Reeves, MD, Principal Investigator — White Clover Wellness and Research Center
Locations (1):
- White Clover Wellness and Research Center, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giuliani A, Fernandez M, Farinelli M, Baratto L, Capra R, Rovetta G, Monteforte P, Giardino L, Calza L. Very low level laser therapy attenuates edema and pain in experimental models. Int J Tissue React. 2004;26(1-2):29-37. PMID 15573690
- [Background] Xu Y, Lin Y, Gao S. Study on the selection of laser wavelengths in the intravascular low-level laser irradiation therapy. Lasers Med Sci. 2015 May;30(4):1373-6. doi: 10.1007/s10103-015-1732-7. Epub 2015 Mar 24. PMID 25800533
- [Background] Martin W. Robert F. Furchgott, Nobel laureate (1916-2009)--a personal reflection. Br J Pharmacol. 2009 Oct;158(3):633-7. doi: 10.1111/j.1476-5381.2009.00418.x. Epub 2009 Aug 13. PMID 19681890
- [Background] Ehrreich SJ, Furchgott RF. Relaxation of mammalian smooth muscles by visible and ultraviolet radiation. Nature. 1968 May 18;218(5142):682-4. doi: 10.1038/218682a0. No abstract available. PMID 5655961
- [Background] Hegedus B, Viharos L, Gervain M, Galfi M. The effect of low-level laser in knee osteoarthritis: a double-blind, randomized, placebo-controlled trial. Photomed Laser Surg. 2009 Aug;27(4):577-84. doi: 10.1089/pho.2008.2297. PMID 19530911
- [Background] Mi XQ, Chen JY, Cen Y, Liang ZJ, Zhou LW. A comparative study of 632.8 and 532 nm laser irradiation on some rheological factors in human blood in vitro. J Photochem Photobiol B. 2004 Mar 19;74(1):7-12. doi: 10.1016/j.jphotobiol.2004.01.003. PMID 15043841
- [Background] Fukuzaki Y, Sugawara H, Yamanoha B, Kogure S. 532 nm low-power laser irradiation recovers gamma-secretase inhibitor-mediated cell growth suppression and promotes cell proliferation via Akt signaling. PLoS One. 2013 Aug 7;8(8):e70737. doi: 10.1371/journal.pone.0070737. eCollection 2013. PMID 23950991
- [Background] Pereira AN, Eduardo Cde P, Matson E, Marques MM. Effect of low-power laser irradiation on cell growth and procollagen synthesis of cultured fibroblasts. Lasers Surg Med. 2002;31(4):263-7. doi: 10.1002/lsm.10107. PMID 12355572
- [Background] Rodrigo SM, Cunha A, Pozza DH, Blaya DS, Moraes JF, Weber JB, de Oliveira MG. Analysis of the systemic effect of red and infrared laser therapy on wound repair. Photomed Laser Surg. 2009 Dec;27(6):929-35. doi: 10.1089/pho.2008.2306. PMID 19708798
- [Background] Lopes NN, Plapler H, Lalla RV, Chavantes MC, Yoshimura EM, da Silva MA, Alves MT. Effects of low-level laser therapy on collagen expression and neutrophil infiltrate in 5-fluorouracil-induced oral mucositis in hamsters. Lasers Surg Med. 2010 Aug;42(6):546-52. doi: 10.1002/lsm.20920. PMID 20662031
- [Background] Yu W, Naim JO, Lanzafame RJ. Effects of photostimulation on wound healing in diabetic mice. Lasers Surg Med. 1997;20(1):56-63. doi: 10.1002/(sici)1096-9101(1997)20:13.0.co;2-y. PMID 9041509
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Medrado AR, Pugliese LS, Reis SR, Andrade ZA. Influence of low level laser therapy on wound healing and its biological action upon myofibroblasts. Lasers Surg Med. 2003;32(3):239-44. doi: 10.1002/lsm.10126. PMID 12605432
- [Background] Hwang MH, Shin JH, Kim KS, Yoo CM, Jo GE, Kim JH, Choi H. Low level light therapy modulates inflammatory mediators secreted by human annulus fibrosus cells during intervertebral disc degeneration in vitro. Photochem Photobiol. 2015 Mar-Apr;91(2):403-10. doi: 10.1111/php.12415. Epub 2015 Jan 26. PMID 25557915
- [Background] Lim W, Choi H, Kim J, Kim S, Jeon S, Zheng H, Kim D, Ko Y, Kim D, Sohn H, Kim O. Anti-inflammatory effect of 635 nm irradiations on in vitro direct/indirect irradiation model. J Oral Pathol Med. 2015 Feb;44(2):94-102. doi: 10.1111/jop.12204. Epub 2014 Jul 28. PMID 25066944
- [Background] Mizutani K, Musya Y, Wakae K, Kobayashi T, Tobe M, Taira K, Harada T. A clinical study on serum prostaglandin E2 with low-level laser therapy. Photomed Laser Surg. 2004 Dec;22(6):537-9. doi: 10.1089/pho.2004.22.537. PMID 15684758
- [Background] Jackson A. Performing peripheral intravenous cannulation. Prof Nurse. 1997 Oct;13(1):21-5. PMID 9393049
- [Background] Blum A, Ovadia M, Rosen G, Simsolo C. Immediate recovery of an "ischemic stroke" following treatment with intravenous thiamine (vitamin B1). Isr Med Assoc J. 2014 Aug;16(8):518-9. No abstract available. PMID 25269348
- [Background] Patil S, Joshi M, Pathak S, Sharma S, Patravale V. Intravenous beta-artemether formulation (ARM NLC) as a superior alternative to commercial artesunate formulation. J Antimicrob Chemother. 2012 Nov;67(11):2713-6. doi: 10.1093/jac/dks293. Epub 2012 Aug 16. PMID 22899802
- [Background] Craven DE, Hudcova J, Lei Y. Ventilator-associated tracheobronchitis: pre-emptive, appropriate antibiotic therapy recommended. Crit Care. 2014 Nov 19;18(6):627. doi: 10.1186/s13054-014-0627-5. PMID 25672436
- [Background] Miller VS, Bates GP. Hydration, hydration, hydration. Ann Occup Hyg. 2010 Mar;54(2):134-6. doi: 10.1093/annhyg/mep091. Epub 2009 Dec 15. PMID 20008893
- [Background] Wendt D, van Loon LJ, Lichtenbelt WD. Thermoregulation during exercise in the heat: strategies for maintaining health and performance. Sports Med. 2007;37(8):669-82. doi: 10.2165/00007256-200737080-00002. PMID 17645370
- [Background] Knowles JR. Enzyme-catalyzed phosphoryl transfer reactions. Annu Rev Biochem. 1980;49:877-919. doi: 10.1146/annurev.bi.49.070180.004305. No abstract available. PMID 6250450
- [Background] Huang YY, Chen AC, Carroll JD, Hamblin MR. Biphasic dose response in low level light therapy. Dose Response. 2009 Sep 1;7(4):358-83. doi: 10.2203/dose-response.09-027.Hamblin. PMID 20011653
- [Background] Karu TI. Mitochondrial signaling in mammalian cells activated by red and near-IR radiation. Photochem Photobiol. 2008 Sep-Oct;84(5):1091-9. doi: 10.1111/j.1751-1097.2008.00394.x. Epub 2008 Jul 18. PMID 18651871
- [Background] Karu T. Photobiology of low-power laser effects. Health Phys. 1989 May;56(5):691-704. doi: 10.1097/00004032-198905000-00015. PMID 2651364
- [Background] Brunori M, Giuffre A, Sarti P. Cytochrome c oxidase, ligands and electrons. J Inorg Biochem. 2005 Jan;99(1):324-36. doi: 10.1016/j.jinorgbio.2004.10.011. PMID 15598510
- [Background] Passarella S, Casamassima E, Molinari S, Pastore D, Quagliariello E, Catalano IM, Cingolani A. Increase of proton electrochemical potential and ATP synthesis in rat liver mitochondria irradiated in vitro by helium-neon laser. FEBS Lett. 1984 Sep 17;175(1):95-9. doi: 10.1016/0014-5793(84)80577-3. No abstract available. PMID 6479342
- [Background] Karu TI, Piatibrat LV, Kalendo GS, Serebriakov NG. [Changes in the amount of ATP in HeLa cells under the action of He-Ne laser radiation]. Biull Eksp Biol Med. 1993 Jun;115(6):617-8. Russian. PMID 8374142
- [Background] Wong-Riley MT, Bai X, Buchmann E, Whelan HT. Light-emitting diode treatment reverses the effect of TTX on cytochrome oxidase in neurons. Neuroreport. 2001 Oct 8;12(14):3033-7. doi: 10.1097/00001756-200110080-00011. PMID 11568632
- [Background] Pastore D, Greco M, Passarella S. Specific helium-neon laser sensitivity of the purified cytochrome c oxidase. Int J Radiat Biol. 2000 Jun;76(6):863-70. doi: 10.1080/09553000050029020. PMID 10902741
- [Background] Eells JT, Wong-Riley MT, VerHoeve J, Henry M, Buchman EV, Kane MP, Gould LJ, Das R, Jett M, Hodgson BD, Margolis D, Whelan HT. Mitochondrial signal transduction in accelerated wound and retinal healing by near-infrared light therapy. Mitochondrion. 2004 Sep;4(5-6):559-67. doi: 10.1016/j.mito.2004.07.033. PMID 16120414
- [Background] Castro-e-Silva T, Castro-e-Silva O, Kurachi C, Ferreira J, Zucoloto S, Bagnato VS. The use of light-emitting diodes to stimulate mitochondrial function and liver regeneration of partially hepatectomized rats. Braz J Med Biol Res. 2007 Aug;40(8):1065-9. doi: 10.1590/s0100-879x2007000800006. PMID 17665042
- [Background] Wong-Riley MT, Liang HL, Eells JT, Chance B, Henry MM, Buchmann E, Kane M, Whelan HT. Photobiomodulation directly benefits primary neurons functionally inactivated by toxins: role of cytochrome c oxidase. J Biol Chem. 2005 Feb 11;280(6):4761-71. doi: 10.1074/jbc.M409650200. Epub 2004 Nov 22. PMID 15557336
- [Background] Kassak P, Przygodzki T, Habodaszova D, Bryszewska M, Sikurova L. Mitochondrial alterations induced by 532 nm laser irradiation. Gen Physiol Biophys. 2005 Jun;24(2):209-20. PMID 16118473
- [Background] Kassak P, Sikurova L, Kvasnicka P, Bryszewska M. The response of Na+/K+ -ATPase of human erythrocytes to green laser light treatment. Physiol Res. 2006;55(2):189-194. doi: 10.33549/physiolres.930711. Epub 2005 May 24. PMID 15910177
- [Background] Muller-Enoch D. Blue light mediated photoreduction of the flavoprotein NADPH-cytochrome P450 reductase. A Forster-type energy transfer. Z Naturforsch C J Biosci. 1997 Sep-Oct;52(9-10):605-14. doi: 10.1515/znc-1997-9-1007. PMID 9373993
- [Background] Leal-Junior EC, Vanin AA, Miranda EF, de Carvalho Pde T, Dal Corso S, Bjordal JM. Effect of phototherapy (low-level laser therapy and light-emitting diode therapy) on exercise performance and markers of exercise recovery: a systematic review with meta-analysis. Lasers Med Sci. 2015 Feb;30(2):925-39. doi: 10.1007/s10103-013-1465-4. Epub 2013 Nov 19. PMID 24249354
- [Background] Brown GC. Nitric oxide regulates mitochondrial respiration and cell functions by inhibiting cytochrome oxidase. FEBS Lett. 1995 Aug 7;369(2-3):136-9. doi: 10.1016/0014-5793(95)00763-y. PMID 7649245
- [Background] Lane N. Cell biology: power games. Nature. 2006 Oct 26;443(7114):901-3. doi: 10.1038/443901a. No abstract available. PMID 17066004
- [Background] Storz P. Mitochondrial ROS--radical detoxification, mediated by protein kinase D. Trends Cell Biol. 2007 Jan;17(1):13-8. doi: 10.1016/j.tcb.2006.11.003. Epub 2006 Nov 28. PMID 17126550
- [Background] Karu T. Primary and secondary mechanisms of action of visible to near-IR radiation on cells. J Photochem Photobiol B. 1999 Mar;49(1):1-17. doi: 10.1016/S1011-1344(98)00219-X. PMID 10365442
- [Background] Alexandratou E, Yova D, Handris P, Kletsas D, Loukas S. Human fibroblast alterations induced by low power laser irradiation at the single cell level using confocal microscopy. Photochem Photobiol Sci. 2002 Aug;1(8):547-52. doi: 10.1039/b110213n. PMID 12659495
- [Background] Chen AC, Arany PR, Huang YY, Tomkinson EM, Sharma SK, Kharkwal GB, Saleem T, Mooney D, Yull FE, Blackwell TS, Hamblin MR. Low-level laser therapy activates NF-kB via generation of reactive oxygen species in mouse embryonic fibroblasts. PLoS One. 2011;6(7):e22453. doi: 10.1371/journal.pone.0022453. Epub 2011 Jul 21. PMID 21814580
- [Background] Grossman N, Schneid N, Reuveni H, Halevy S, Lubart R. 780 nm low power diode laser irradiation stimulates proliferation of keratinocyte cultures: involvement of reactive oxygen species. Lasers Surg Med. 1998;22(4):212-8. doi: 10.1002/(sici)1096-9101(1998)22:43.0.co;2-s. PMID 9603282
- [Background] Valencia A, Kochevar IE. Nox1-based NADPH oxidase is the major source of UVA-induced reactive oxygen species in human keratinocytes. J Invest Dermatol. 2008 Jan;128(1):214-22. doi: 10.1038/sj.jid.5700960. Epub 2007 Jul 5. PMID 17611574
- [Background] Lavi R, Shainberg A, Friedmann H, Shneyvays V, Rickover O, Eichler M, Kaplan D, Lubart R. Low energy visible light induces reactive oxygen species generation and stimulates an increase of intracellular calcium concentration in cardiac cells. J Biol Chem. 2003 Oct 17;278(42):40917-22. doi: 10.1074/jbc.M303034200. Epub 2003 Jul 7. PMID 12851407
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Background] Aimbire F, Albertini R, Pacheco MT, Castro-Faria-Neto HC, Leonardo PS, Iversen VV, Lopes-Martins RA, Bjordal JM. Low-level laser therapy induces dose-dependent reduction of TNFalpha levels in acute inflammation. Photomed Laser Surg. 2006 Feb;24(1):33-7. doi: 10.1089/pho.2006.24.33. PMID 16503786
- [Background] Piva JA, Abreu EM, Silva Vdos S, Nicolau RA. Effect of low-level laser therapy on the initial stages of tissue repair: basic principles. An Bras Dermatol. 2011 Sep-Oct;86(5):947-54. doi: 10.1590/s0365-05962011000500013. No abstract available. English, Portuguese. PMID 22147035
- [Background] Ferreira DM, Zangaro RA, Villaverde AB, Cury Y, Frigo L, Picolo G, Longo I, Barbosa DG. Analgesic effect of He-Ne (632.8 nm) low-level laser therapy on acute inflammatory pain. Photomed Laser Surg. 2005 Apr;23(2):177-81. doi: 10.1089/pho.2005.23.177. PMID 15910182
- [Background] Bjordal JM, Lopes-Martins RA, Iversen VV. A randomised, placebo controlled trial of low level laser therapy for activated Achilles tendinitis with microdialysis measurement of peritendinous prostaglandin E2 concentrations. Br J Sports Med. 2006 Jan;40(1):76-80; discussion 76-80. doi: 10.1136/bjsm.2005.020842. PMID 16371497
- [Background] Zhevago NA, Samoilova KA. Pro- and anti-inflammatory cytokine content in human peripheral blood after its transcutaneous (in vivo) and direct (in vitro) irradiation with polychromatic visible and infrared light. Photomed Laser Surg. 2006 Apr;24(2):129-39. doi: 10.1089/pho.2006.24.129. PMID 16706691
- [Background] Bjordal JM, Couppe C, Chow RT, Tuner J, Ljunggren EA. A systematic review of low level laser therapy with location-specific doses for pain from chronic joint disorders. Aust J Physiother. 2003;49(2):107-16. doi: 10.1016/s0004-9514(14)60127-6. PMID 12775206
- [Background] Wilson, J. (2006) Preventing infection associated with intravascular therapy In: Infection Control in Clinical Practice 3rd ed. Baillière Tindall London 199-213.
- [Background] Fu XJ, Peng YB, Hu YP, Shi YZ, Yao M, Zhang X. NADPH oxidase 1 and its derived reactive oxygen species mediated tissue injury and repair. Oxid Med Cell Longev. 2014;2014:282854. doi: 10.1155/2014/282854. Epub 2014 Jan 19. PMID 24669283
- [Background] Hamblin MR, Tatiana ND. Mechanisms of low level light therapy. Proc. SPIE 6140, Mechanisms for Low-Light Therapy, 614001 (February 10, 2006)
- [Background] Alves AC, Vieira R, Leal-Junior E, dos Santos S, Ligeiro AP, Albertini R, Junior J, de Carvalho P. Effect of low-level laser therapy on the expression of inflammatory mediators and on neutrophils and macrophages in acute joint inflammation. Arthritis Res Ther. 2013;15(5):R116. doi: 10.1186/ar4296. PMID 24028507
- [Background] Bjordal JM, Johnson MI, Iversen V, Aimbire F, Lopes-Martins RA. Low-level laser therapy in acute pain: a systematic review of possible mechanisms of action and clinical effects in randomized placebo-controlled trials. Photomed Laser Surg. 2006 Apr;24(2):158-68. doi: 10.1089/pho.2006.24.158. PMID 16706694
- [Background] Lopes NN, Plapler H, Chavantes MC, Lalla RV, Yoshimura EM, Alves MT. Cyclooxygenase-2 and vascular endothelial growth factor expression in 5-fluorouracil-induced oral mucositis in hamsters: evaluation of two low-intensity laser protocols. Support Care Cancer. 2009 Nov;17(11):1409-15. doi: 10.1007/s00520-009-0603-9. Epub 2009 Feb 22. PMID 19234862
- [Background] de Jesus JF, Spadacci-Morena DD, dos Anjos Rabelo ND, Pinfildi CE, Fukuda TY, Plapler H. Low-level laser therapy in IL-1beta, COX-2, and PGE2 modulation in partially injured Achilles tendon. Lasers Med Sci. 2015 Jan;30(1):153-8. doi: 10.1007/s10103-014-1636-y. Epub 2014 Jul 29. PMID 25070591
- [Background] de Morais NC, Barbosa AM, Vale ML, Villaverde AB, de Lima CJ, Cogo JC, Zamuner SR. Anti-inflammatory effect of low-level laser and light-emitting diode in zymosan-induced arthritis. Photomed Laser Surg. 2010 Apr;28(2):227-32. doi: 10.1089/pho.2008.2422. PMID 19780633
- [Background] Tanno Y, Mahmood A. Liver Repair in Rabbits Using 532 nm Nd:YAG Laser; In Vivo Study. Iraqi J. Laser, Part B, Vol.10, No.1, pp. 25-30 (2011)
- [Background] Vinck EM, Cagnie BJ, Cornelissen MJ, Declercq HA, Cambier DC. Green light emitting diode irradiation enhances fibroblast growth impaired by high glucose level. Photomed Laser Surg. 2005 Apr;23(2):167-71. doi: 10.1089/pho.2005.23.167. PMID 15910180
- [Background] Schwengel RH, Gregory KW, Hearne SE, Scott HJ, Beauman GJ, Mergner WJ, Caplin JL, Ziskind AA. Characterization of pulsed-dye laser-mediated vasodilatation in a rabbit femoral artery model of vasoconstriction. Lasers Surg Med. 1993;13(3):284-95. doi: 10.1002/lsm.1900130305. PMID 8515668
- [Background] Xiaosen L, Ni Xiaowu L, Jian HA, Liu Xiaoran X, Jiangying SJ. (2002) Influence of He-Ne laser on oxygen dissociation of erythrocyte. J J Optoelectron•Laser 13(4):413-415
- [Background] Luo X, Ni X, Lu J, He A, Liu X, Liu J, Li L (2001) Influence of Laser Irradiation on the Process of Blood Oxygenation. J J Optoelectron•Laser 12(11):1196-1198